CLINICAL TRIAL: NCT04585880
Title: Remote Monitoring and Virtual Collaborative Care For Hypertension Control To Prevent Cognitive Decline: Phase I
Brief Title: Remote Monitoring and Virtual Collaborative Care For Hypertension Control To Prevent Cognitive Decline
Acronym: vCCC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Jeff Burns, MD, Co-Director Alzheimer's Disease Center, University of Kansas Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY146086; 1R61AG068483-01 (NIH)
Record Dates: First submitted 2020-09-30; First posted 2020-10-14 (Actual); Last update posted 2021-07-09 (Actual); Status verified 2021-07

CONDITIONS: Hypertension; Cognitive Decline
Keywords: Hypertension; Cognitive Decline; Mild Cognitive Decline; Memory Loss; Memory Disorders; Memory Impairment; Blood Pressure; Blood Pressure, High
MeSH Terms: conditions — Hypertension; Cognitive Dysfunction; Memory Disorders

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Collaborative Care Clinic (Experimental): The Virtual Collaborative Care Clinic arm participants use a home blood pressure monitor and routine blood pressure measurements will be uploaded to a dashboard monitored by clinical pharmacists. Blood pressure will be managed aggressively by the clinical pharmacists in coordination with Primary Care Physicians.
  Interventions: Other: Virtual Collaborative Care Clinic
- Control Intervention (No Intervention): The control intervention will consist of providing the participant with educational material and a home blood pressure monitor. The patients in the control group will not have support from Virtual Collaborative Care Clinic pharmacists. Routine blood pressure measures using their device will not be collected via the dashboard and will not be available for pharmacist review. Participants will continue to see their physicians for their usual care for blood pressure management.

INTERVENTIONS:
Other: Virtual Collaborative Care Clinic — The vCCC will operate under a collaborative care agreement with the Primary Care Physicians as an extension (and not a replacement) of their care. Trained clinical pharmacists will monitor blood pressure and prescribe and adjust medications under the license of, and in communication with, the patient's Primary Care Physician. As part of the Primary Care Physician's team and per Primary Care Physician's directions, the pharmacists may coordinate blood pressure management with other clinicians such as cardiologists or nephrologists co-managing patients blood pressure.
  Arms: Virtual Collaborative Care Clinic

SUMMARY:
This purpose of this study is to examine an aggressive method of blood pressure control that involves home blood pressure monitoring and management of medications by a team of clinical pharmacists in coordination with a primary care physician.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 and older
* Active patient in participating primary care clinic
* Access to compatible "smartphone" or device (i.e., Android, Kindle or Apple with internet connectivity)
* Elevated blood pressure as defined by:

Systolic Blood Pressure >140 at current visit AND documented history of hypertension OR Systolic Blood Pressure > 140 at current visit and at another visit in last 18 months OR Systolic Blood Pressure >160 at current visit

* Sufficiently fluent in English to participate in study procedures
* Adequate vision and hearing to complete study procedures

Exclusion Criteria:

* Clinically significant illness that may affect safety or completion per their treating Primary Care Physician or study physician
* End stage renal disease on dialysis
* Chronic active disease with expected life expectancy < 2 years as determined by the study team

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 33 (Actual)
Dates: Start 2020-10-20 (Actual); Primary Completion 2021-07-02 (Actual); Study Completion 2021-07-02 (Actual)

PRIMARY OUTCOMES:
Feasibility of system wide adoptability as assessed by survey responses | Baseline
  Primary Care Physicians and vCCC Pharmacists will be asked for feedback on feasibility of implementation via a survey. The vCCC pharmacists and PCPs will be surveyed to assess feasibility and changing views of feasibility. Brief, validated scales will be delivered via email (REDCap surveys) to assess the construct of feasibility.
Feasibility of system wide adoptability as assessed by survey responses | 3 Months Post Baseline
  Primary Care Physicians and vCCC Pharmacists will be asked for feedback on feasibility of implementation via a survey. The vCCC pharmacists and PCPs will be surveyed to assess feasibility and changing views of feasibility. Brief, validated scales will be delivered via email (REDCap surveys) to assess the construct of feasibility.
Feasibility of system wide adoptability as assessed by Physician Advisory Board meetings discussion | Through study completion, an average of 9 months
  Members of the Physician Advisory Board will be asked for feedback on system wide adoptability during the monthly Physician Advisory Board meetings. The meetings will be recorded and summarized.
Feasibility of system wide adoptability as assessed by vCCC Pharmacist Interviews | Up to 2 months Post Baseline
  Virtual Collaborative Care Clinic Pharmacists will be asked for feedback on feasibility of system wide adoption. We will conduct one-time semi-structured qualitative interviews with the Virtual Collaborative Care Clinic pharmacists. The Virtual Collaborative Care Clinic pharmacist will be interviewed to assess implementation factors including the auto-referral process and open-ended questions on the process and suggestions for improvement.
Replicability to other health systems as assessed by survey responses | Baseline
  Primary Care Physicians and vCCC Pharmacists will be asked for feedback on replicability to other health systems via a survey. Brief, validated scales will be delivered via email (REDCap surveys) to assess the construct of replicability to other health systems.
Replicability to other health systems as assessed by survey responses | 3 Months Post Baseline
  Primary Care Physicians and vCCC Pharmacists will be asked for feedback on replicability to other health systems via a survey. Brief, validated scales will be delivered via email (REDCap surveys) to assess the construct of replicability to other health systems.
Replicability to other health systems as assessed by Physician Advisory Board meetings discussion | Through study completion, an average of 9 months
  Members of the Physician Advisory Board will be asked for feedback on replicability to other health systems during the monthly Physician Advisory Board meetings. The meetings will be recorded and summarized.
Replicability to other health systems as assessed by vCCC Pharmacist Interviews | Up to 2 months Post Baseline
  vCCC Pharmacists will be asked for feedback on replicability to other health systems. We will conduct one-time semi-structured qualitative interviews including open-ended questions.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Burns, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No